CLINICAL TRIAL: NCT02012049
Title: Bioequivalence Test for Risperdal OD Tab. 2mg of Janssen Korea
Brief Title: Bioequivalence Test for Risperdal 2mg of Janssen Korea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR016576; RISSCH1015 (Other: Janssen Korea, Ltd., Korea); RIS-KOR-1083 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2013-12-10; First posted 2013-12-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: Healthy; Risperdal OD; Risperdal Quicklet; Korea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risperdal OD / Risperdal Quicklet (Experimental): Risperdal OD (investigational drug) + Risperdal Quicklet (control drug)
  Interventions: Drug: Risperdal OD Tab. 2mg; Drug: Risperdal Quicklet Tab. 2mg
- Risperdal Quicklet / Risperdal OD (Experimental): Risperdal Quicklet (control drug) + Risperdal OD (investigational drug)
  Interventions: Drug: Risperdal OD Tab. 2mg; Drug: Risperdal Quicklet Tab. 2mg

INTERVENTIONS:
Drug: Risperdal OD Tab. 2mg — 1 tablet Risperdal OD 2 mg administered orally.
Drug: Risperdal Quicklet Tab. 2mg — 1 tablet Risperdal Quicklet Tab. 2mg administered orally.

SUMMARY:
The purpose of this study was to conduct the bioequivalence (biological equivalence of two preparations of a drug) test in healthy adults with "Risperdal OD Tab. 2mg" of Janssen Korea as the investigational drug and "Risperdal Quicklet Tab. 2mg" as the control drug.

DETAILED DESCRIPTION:
This was a randomized (the study drug is assigned by chance) and open labeled (all people know the identity of the intervention) study. All participants were hospitalized in research rooms and were subsequently restricted in exercise, eating, drinking, smoking and xanthine-beverages until the end of blood collection. Water was allowed to be taken until one hour before drug administration. Participants were randomly assigned into two groups, one group receiving Risperdal OD (investigational drug), and one group receiving Risperdal Quicklet (control drug). On the day of testing, blood was collected from all participants to provide baseline measurements. Subsequently, the study drug was orally administered to the participants, followed by blood collection of a total of 13 time points, up to 24 hours. After the blood collection was finished, participants were discharged after receiving proper guidance and being examined by a psychologist. Following a wash-out period (period when receiving no intervention) of one week, participants were hospitalized once more and crossed over to receive the study drugs following the same procedure above described. The approximate study duration (including the drug administration days and wash-out period) was approximately 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Korean participants weighing more than 50kg and within 20% normal lean body weight (standard weight)
* Participant without congenital or chronic diseases and with no symptoms or findings as a result of internal examination
* Participant who was deemed appropriate as a result of inquiry, blood pressure, physical examination, electrocardiogram, blood and urinalysis, etc., within 28 days prior to the first administration of the investigational drug according to the protocol
* Female participant who was confirmed as non-pregnant through urine test during health examination

Exclusion Criteria:

* Participant who had a history of disease related to cardiac, respiratory, hepatic, renal, gastrointestinal or nervous system, or cardiac infarction, stroke, hypertension, arrhythmia, coronary artery disease, or neuropsychiatric diseases that could affect drug absorption, distribution, metabolism and excretion or could be risk factors when taking drugs used for the clinical trial, a history of gastrointestinal surgery except appendectomy or herniotomy, or who currently had abnormality in inquiry or physical examination
* Participant who showed symptoms that were suspected as acute disease within 14 days from the first administration of the investigational drug
* Participant with allergic disease requiring treatment
* Participant who had a history of being hypersensitive to drugs or food
* Patient who had hepatitis B antigen or who showed hepatitis C positive antigen

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of Risperidone | Up to 24 hours postdose

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety | Approximately 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea